CLINICAL TRIAL: NCT01807429
Title: Comparing Low Dose IV Ketamine-midazolam Versus IV Morphine Regarding ED Pain Control in Patients Sustaining Closed Limb Fracture(s)
Brief Title: Is Analgesic Effect of Low Dose Ketamine-midazolam the Same as Morphine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Mehdi Nasr Isfahani, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 390284
Record Dates: First submitted 2013-02-21; First posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Closed Multiple Fractures of Upper and Lower Limbs
Keywords: Ketamine,; Midazolam,; Morphine,; visual analogue score
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine-midazolam (Experimental): 300 to 500 mcg/kg ketamine plus 0.03 mg/kg midazolam
  Interventions: Drug: Ketamine-midazolam
- Morphine (Active Comparator): 0.05 to 0.1 mg/kg morphine
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine-midazolam — Ketamine 300-500mcg/kg plus midazolam 0.03 mg/kg once.
  Other Names: Ketaral
  Arms: Ketamine-midazolam
Drug: Morphine — morphine 0.05 mg/kg
  Other Names: Avinza
  Arms: Morphine

SUMMARY:
the investigators assessed the effects of low-dose IV ketamine-midazolam versus morphine on pain control in trauma patients with closed limb fracture(s); and also compared the incidence of adverse events (mainly cardio pulmonary ) between two groups.

DETAILED DESCRIPTION:
this prospective, single blind, noninferiority trial randomized consecutive ED patients aged 18 to 60 years to two groups: receiving either 300-500 mcg ketamine plus 0.03 mg midazolam, or 0.05 to 0.1 mg morphine. Visual analogue score and adverse events were carefully verified during an interval of 30 minutes.

Two hundreds, thirty six patients were selected, among whom were 207 males (87.3%), and 29 females (12.2%). The average age was 29±2, with extremes of 60 years and 18 years.the patients were divided into two groups: G1: 116 patients receiving ketamine-midazolam and G2: 120 patients receiving morphine alone.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 60 years
2. Patients with closed limb fracture(s)
3. VAS score of at least 6

Exclusion Criteria:

1. Acute pulmonary infection
2. Previous coronary artery diseases,ACS,congestive heart failure,
3. suspected aortic dissection
4. History of uncontrolled hypertention or blood pressure > 140/90mmHg
5. Brain injury with focal neurological deficit or loss of consciousness
6. Central nervous system mass lesion,hydrocephalus, or other states with increased intracranial pressure
7. Glaucoma and acute globe injury
8. History of porphyria
9. Previous hyperthyroidism or thyroid hormone replacement
10. Pregnancy or laction
11. Major psychiatric disorder
12. Previous allergic reaction to the agents administered in the study
13. Patient declined to provide written informed conse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
VAPS | 30 minutes
  the pain score was verified at the outset and every 10 minutes after administration of analgesics.

SECONDARY OUTCOMES:
HR,RR,SPO2,BP | 30 minutes
  the variables were assessed for an interval of 30 minutes.

OTHER OUTCOMES:
adverse drug effects | 30 minutes
  the patients were closely observed for any drug induced adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Omid Ahmadi, professor, Study Director — Isfahan University of Medical Sciences